CLINICAL TRIAL: NCT04141501
Title: Phase II, Randomized, Double Blind, Placebo Controlled, Parallel Group, Single Center Study of Psilocybin Efficacy and Mechanism in Alcohol Use Disorder
Brief Title: Clinical and Mechanistic Effects of Psilocybin in Alcohol Addicted Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Schweizerischer Nationalfonds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PsiAlc133
Record Dates: First submitted 2019-10-03; First posted 2019-10-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Use Disorder
Keywords: Alcoholism; Psilocybin; Psychedelics; clinical efficacy; autobiographical memory; cue-reactivity exposure; placebo-controlled; proof-of-concept
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Phase II, randomized, double blind, placebo controlled, parallel group, single center study
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Placebo (Placebo Comparator): 30 Patients will receive placebo
  Interventions: Drug: Placebo oral capsule
- Intervention: Psilocybin (Active Comparator): 30 Patients will receive psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — single dose of psilocybin (25mg). orally in form of a capsule
  Arms: Intervention: Psilocybin
Drug: Placebo oral capsule — single dose of mannitol (100%)
  Arms: Control: Placebo

SUMMARY:
Effects of serotonin 2A/1A receptor stimulation by psilocybin on alcohol addicted patients: a randomized double-blind placebo-controlled study

DETAILED DESCRIPTION:
Two billion people globally consume alcohol, leading in 2016 to 2.8 million deaths (5.2% of all deaths) and 99.2 million Disability Adjusted Life Years (DALYs) lost (4.2% of all DALYs). Of all the diseases, conditions, and injuries attributable to alcohol use, alcohol use disorders (AUDs) create the largest health burden globally. However, approved pharmacological treatments for alcoholism are limited in their effectiveness. A recent proof of- concept study testing psilocybin in ten alcohol dependent patients provides encouraging efficacy results and safety data. The investigators, therefore, propose to test the efficacy of psilocybin for treating alcohol use disorder and study its underlying neurobiological mechanisms in a randomized, placebo controlled, double blind study. To evaluate effects of psilocybin on alcohol use behaviour, clinical symptoms, neurocognitive and emotional measures in patients with alcohol use disorder.

The present clinical trial aims at investigation the clinical and mechanistic effects of Psilocybin in Alcohol Addicted Patients.

Patients with alcohol use disorder who have undergone withdrawal treatment within the last 6 weeks will be investigated in a single-centre, double-blind, placebo-controlled, parallel-group design clinical trial contrasting the acute and persisting effects of psilocybin to those of placebo. Patients will be randomly assigned to psilocybin or placebo group with a 1:1 allocation ratio. The study comprises a total of 6 visits during 6 weeks and two follow-up online surveys (3 and 6 months after treatment). In addition, two follow-up surveys that can be completed from home will guarantee monitoring of long-lasting changes in symptomology and ensure all potential side-effects can be captured. On the treatment visit, a single dose of psilocybin (25mg) or placebo will be administered. Patients will be monitored until all effects have worn off.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Right-handedness according to Oldfield (1971) perfomed during the telephone screening, laterality index ≥ 0.2
* DSM-IV-diagnosis of alcohol use disorder (based on clinical assessment and confirmed by the SCID Interview)
* Having undergone withdrawal treatment from alcohol use or have stopped consuming alcohol within 6 weeks prior to enrolment in the study
* Drug free from any psychotropic and serotonergic medication for at least five days before administration of the study drug or placebo
* No alcohol use between withdrawal treatment and administration of study drug or placebo
* Good physical health with no unstable medical conditions, as determined by medical history, physical examination, routine blood labs, electrocardiogram, urine analysis, and urine toxicology
* Normal level of language comprehension (German or Swiss-German)
* Willing to refrain from drinking caffeinated drinks during the testing days and from consuming psychoactive substances after enrolling in the study and for the remainder of the study
* Women of childbearing potential must be using an effective, established method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices. Note: female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Have a family member or friend who can pick them up and stay with them overnight after the psilocybin administration sessions (driving is forbidden at drug treatment days)
* No further medication is allowed until visit 6, except for emergencies

Exclusion Criteria:

* Allergy, hypersensitivity, or other adverse reaction to previous use of psilocybin or other hallucinogens
* uncorrected Hypertension (assessed at screening day: higher than 139 systolic and 89 diastolic)
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases (Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential)
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Lifetime history of bipolar disorder (I, II, not otherwise specified) Lifetime history of schizophrenia, schizoaffective disorder, or psychosis not otherwise specified
* History of DSM-IV drug dependence other than alcohol (except for caffeine or nicotine) within two months prior to enrolment
* Comorbid Axis I anxiety and depression disorders diagnoses as well as post-traumatic stress disorder will be permitted if they do not require current treatment
* Family history of schizophrenia or schizoaffective disorder, or bipolar disorder type 1 (first or second degree relatives)
* Violent behaviour within last 2 years or history of suicidal behaviour
* Lifetime history of hallucinogen use on more than 10 occasions within last 10 years
* Getting psychotherapeutic or psychological treatment from third parties during the study is forbidden
* Abnormal electrocardiogram
* Any unstable illness as determined by history or laboratory tests
* BMI <17 or >30
* Uncorrected hypo- or hyperthyroidism
* Contraindications to magnetic resonance imaging (MRI safety form)
* During the study, new use or dose changes of already existing concomitant medication without prior informing the investigators is forbidden
* High risk of adverse emotional or behavioural reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behaviour, serious current stressors, lack of meaningful social support)
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Taking medications that are known to modulate uridine diphosphate glucuronosyltransferase enzyme
* Inhibitors of UGT1A9 and 1A10 should be discontinued at least five half-lives prior to the administration of psilocybin
* Monoamine oxidase and aldehyde or alcohol dehydrogenase inhibitors should be discontinued at least 5 half-lives prior to the dose of psilocybin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Changes in Time-Line Follow-Back | every day from baseline until 6 months after the intervention (primary endpoint: 4 weeks after administration, follow-up period 6 months)
  measures changes of the alcohol use behavior over time.The Time-Line Follow-Back questionnaire assesses the standard glasses of alcohol consumed in a day. The minimum is no alcohol consumption, with the maximum being an open end. Less alcohol consumption will be the better outcome, whereas more alcohol consumption will be a worse outcome.
  The primary efficacy value will be alcohol use (average of daily standard units of alcohol use between visit 3 and visit 6) between psilocybin administration and visit 6 (four weeks after psilocybin administration)
Relapse using Time-Line Follow-Back | Relapse will be compared between the placebo and psilocybin group in the time period four weeks after visit 3
  Re-instatement of alcohol drinking behaviour > 1 standard drink will be defined as relapse.

SECONDARY OUTCOMES:
Brain | The MRI will be completed at baseline (visit 2, approx. 5 days prior), approx. 90 minutes after the administration of the investigational medicinal product (IMP), and following IMP-administration (approx. 4 weeks later).
  Changes in resting-state fMRI, cue-reactivity task fMRI, autobiographic memory task fMRI and DTI. MRI data will be analysed using general lineal models (GLMs) and psychophysiological interaction models. For these analyses, the generally established methods of controlling for multiple comparisons will be applied.
Empathy | five days before IMP-administration, one day post and approx. 4 weeks post intervention
  Changes in empathy assessed with the Multifaceted Empathy Task
Blood sample: Neural profile analysis | At baseline, approx. five days before intervention
  To investigate the in vitro neuronal profile of psilocybin in alcohol dependent individuals blood cells before psilocybin administration will be differentiated into cortical neurons.
Blood sample: Epigenetic analysis | At baseline (approx. five day before intervention), one day after the IMP-administration, and approx. 4 weeks after the IMP-administration
  Genome-wide genetic analyses will be conducted to investigate association between gene variants and treatment outcomes. Genome-wide changes in epigenetic markers of treatment response will be analysed before and after psilocybin administration
Blood sample: Markers of alcohol use | This will be analysed at screening visit and approx. 4 weeks after the IMP-administration.
  Ethylglucuronid, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and gamma-glutamyltransferase (GGT) will be analysed from blood samples (except for Ethylglucuronid which will be analysed in urine samples) as objective markers of alcohol use. Additionally, cortisol will be analysed.
Alcohol Self-Efficacy Scale | The questionnaire will be completed at screening (visit 1, approx. 14 days prior), baseline (visit 2, approx. 5 days prior), and post IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups)
  The Alcohol Self-Efficacy scale measures an individual's confidence in their ability to resist drinking alcohol in high-risk situations. It consists of 20 items and uses a 5-point Likert scale, with 0 representing "not at all confident" and 4 representing "extremely confident." The minimum score possible is 20, and the maximum score is 100.
  Higher scores indicate greater self-efficacy or confidence in one's ability to resist drinking in high-risk situations, while lower scores indicate lower levels of self-efficacy. The scale can be used to assess an individual's readiness to change their drinking behavior and to identify areas where additional support or intervention may be necessary.
Penn Alcohol Craving Scale | The questionnaire will be completed at screening (visit 1, approx. 14 days prior), baseline (visit 2, approx. 5 days prior), directly before IMP administration, and post IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups)
  The Penn Alcohol Craving Scale is a tool used to assess the intensity of an individual's craving for alcohol. It consists of 5 items, each rated on a 7-point Likert scale ranging from 0 (not at all) to 6 (extremely). The minimum score possible is 0, and the maximum score is 30.
  Higher scores on the Penn Alcohol Craving Scale indicate more intense alcohol cravings, while lower scores indicate lower levels of craving. The scale can be used to monitor the effectiveness of treatments aimed at reducing alcohol craving, as well as to identify triggers for alcohol use and to assess an individual's readiness to change their drinking behavior.
Snaith-Hamilton-Pleasure Scale (SHAPS) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).]
  The Snaith-Hamilton-Pleasure Scale (SHAPS) is a tool used to measure an individual's capacity to experience pleasure in daily life. It consists of 14 items and uses a 4-point Likert scale, with 1 representing "strongly disagree" and 4 representing "strongly agree." The minimum score possible is 14, and the maximum score is 56.
  Higher scores on the SHAPS indicate greater capacity for pleasure, while lower scores may suggest anhedonia, which is a reduced ability to experience pleasure. The scale can be used to assess an individual's emotional well-being and screen for depressive symptoms or other mood disorders. Additionally, the scale may be used to monitor the effectiveness of treatment interventions aimed at improving an individual's ability to experience pleasure in daily life.
Number of Heavy Drinking Days (HDDs) | 4 weeks after administration, and at 6 month follow-up
  HDD was defined as a day with alcohol consumption of five or more standard units for a man and four or more standard units for a woman
Time to Relapse | 4 weeks after administration, and at 6 month follow-up
  The Time to Relapse is the amount of self-reported abstinent days post administration until relapse occurs (relapse is defined as > 1 standard drink).
Emotion-Regulation Questionnaire (ERQ) | The questionnaire will be completed at baseline (approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups)
  The ERQ is a self-report tool measuring an individual's tendency to regulate their emotions in two ways: reappraisal and suppression. The scale range for each subscale is as follows: for the reappraisal subscale, the minimum score is 6 and the maximum score is 42; for the suppression subscale, the minimum score is 4 and the maximum score is 28.
  Higher scores on the reappraisal subscale indicate a greater tendency to regulate emotions by reinterpreting them in a more positive light, while higher scores on the suppression subscale indicate a greater tendency to inhibit the expression of emotions. Lower scores on either subscale suggest a weaker tendency to use that emotion regulation strategy.
Savoring Believes Inventory (SBI) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).]
  The SBI is a self-report tool assessing an individual's beliefs towards savoring positive experiences. It consists of 21 items and uses a 4-point Likert scale, with 1 representing "strongly disagree" and 5 representing "strongly agree." The minimum score possible is 24, and the maximum score is 120.
  Higher scores on the SBI indicate a greater tendency to savor positive experiences, while lower scores suggest a weaker tendency to engage in savoring behaviors.
Temporary Experience of Pleasure Scale (TEPS) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).]
  The TEPS is a self-report tool measuring an individual's capacity to experience pleasure in response to natural rewards. The minimum score possible is 18, and the maximum score is 108.
  The TEPS assesses two dimensions of pleasure: anticipatory pleasure and consummatory pleasure.
  Higher scores on the TEPS indicate a greater capacity to experience pleasure in response to natural rewards, while lower scores suggest a reduced ability to experience pleasure. The scale can be used to assess an individual's emotional well-being and to screen for anhedonia, which is a reduced ability to experience pleasure. Additionally, the scale may be used to monitor the effectiveness of treatment interventions aimed at improving an individual's capacity to experience pleasure. The TEPS has been used in research to investigate the relationship between pleasure and various psychological outcomes, such as depression, substance use disorders, and personality traits.
Quality of Life Scale (QOL) | It will be completed at baseline (approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups)
  The QOL is a self-report tool measuring an individual's subjective evaluation of their overall quality of life. The scale measures multiple domains related to quality of life, including physical health, psychological well-being, social relationships, and environmental factors.
  The scale range for each subscale is as follows: for physical health, the minimum score is 4 and the maximum score is 28; for psychological well-being, the minimum score is 5 and the maximum score is 35; for social relationships, the minimum score is 3 and the maximum score is 21; for environmental factors, the minimum score is 4 and the maximum score is 28. The total score for the QOL ranges from 32 to 168.
  Higher scores on the QOL indicate a better quality of life, while lower scores suggest a poorer quality of life.
Positive and Negative Affect Schedule (PANAS) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).
  PANAS is a questionnaire for measuring positive and negative affect. It consists of two 10-item scales, one measuring positive affect (PA) and one measuring negative affect (NA). Each item is rated on a 5-point scale, ranging from "very slightly or not at all" to "extremely". The scores for the PA and NA scales can be summed separately, with higher scores indicating higher levels of positive or negative affect, respectively. The minimum score for the Positive Affect (PA) scale is 10 (when all 10 items are rated as "very slightly or not at all"). The maximum score for the PA scale is 50 (when all 10 items are rated as "extremely"). The minimum score for the Negative Affect (NA) scale is 10 (when all 10 items are rated as "very slightly or not at all"). The maximum score for the NA scale is 50 (when all 10 items are rated as "extremely").
Stundentagebuch, STEPP/STEPT | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).
  The Stundenbogen are short standardized questionnaires for formative evaluation of psychological counseling. Both questionnaires include 12 items which have to be answered by the patient or client or by the psychotherapist or counselor after a psychotherapy or counseling session. Items are constructed complementarily for therapists and patients and refer to (1) the motivational clarification and development of the patient, (2) the active help for problem-solving by the patient and (3) the therapeutic support experienced by the patient (patient questionnaire) versus that perceived by the therapist (therapist questionnaire). Higher scores over time would indicate a better outcome.
Hopelessness-Scale (HS-scale) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).
  The HS-scale is a self-report tool used to measure an individual's level of hopelessness, pessimism, and negative expectations about the future. It consists of 20 items and uses a true-false response format. The scale range for the HS-scale is from 0 to 20, with higher scores indicating greater levels of hopelessness.
  The HS-scale can be used to assess an individual's level of hopelessness and to identify areas where additional support or intervention may be necessary. It is commonly used in clinical and research settings to study the relationship between hopelessness and various psychological outcomes, such as depression, suicidal ideation, and anxiety. The scale may also be used to monitor the effectiveness of treatment interventions aimed at reducing hopelessness and improving mental health outcomes.
Frankfurt Self-Concept Scale (FSKN) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).
  The Frankfurt Self-Concept Scale (FSKN) is a self-report tool assessing an individual's self-concept or self-image. The FSKN measures multiple dimensions of self-concept, including social self-concept, competence self-concept, and affective self-concept.
  The FSKN assesses an individual's self-concept and identifies areas where additional support or intervention may be necessary. It is commonly used in clinical and research settings to study the relationship between self-concept and various psychological outcomes, such as self-esteem, anxiety, and depression. The scale may also be used to monitor the effectiveness of treatment interventions aimed at improving self-concept and overall well-being. Higher scores indicating a more positive self-concept.
Beck Depression Inventory (BDI) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).
  The BDI measures the severity of depression. It consists of 21 items that assess a range of symptoms associated with depression, such as sadness, guilt, worthlessness, and loss of pleasure. Each item is scored on a four-point scale ranging from 0 to 3, with higher scores indicating greater severity of depression. The scale ranges from "0" indicating the absence of the symptom to "3" indicating the most severe form of the symptoms. The total score on the BDI ranges from 0 to 63, with higher scores indicating greater levels of depression.
Hamilton Anxiety Scale (HAMA) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).]
  The Hamilton Anxiety Scale (HAMA) is a questionnaire for assessing the severity of anxiety symptoms. It consists of 14 items that measure both psychic anxiety (e.g., tension, fear, insomnia) and somatic anxiety (e.g., palpitations, sweating, headaches). Each item is scored on a five-point scale ranging from 0 to 4, with higher scores indicating greater severity of anxiety. On this scale, a score of "0" indicates the absence of the symptom, while a score of "1" indicates mild, "2" moderate, "3" severe, and "4" very severe symptoms. The total score on the HAMA ranges from 0 to 56, with higher scores indicating greater levels of anxiety.
The Stress Questionnaire (CQ) | The questionnaire will be completed at baseline (visit 2, approx. 5 days prior), and following IMP administration (1, approx. 14, approx. 28 days post-treatment and follow-ups).]
  The CQ is 7-item self-report scale that measures potential stressors, the burden it elicits and the progress done regarding this issue. It is adapted from the Stress & Coping Inventory. The questionnaire is used to measure a person's level of stress and their ability to manage and cope with it.
Drinker Inventory of Consequences (DrInc) | The questionnaire will be completed at screening (visit 1, approx. 14 days prior to the IMP-administration), and following IMP administration (approx. 28 days post-treatment and follow-ups)
  The "Drinker Inventory of Consequences (DrInc)" is a self-report inventory that measures the negative consequences associated with alcohol use. It consists of 50 items that assess 5 domains of consequences: physical, interpersonal, intrapersonal, impulse control, and social responsibility. The items ask about the frequency and severity of negative consequences experienced due to alcohol use. The DrInc uses a Likert scale, where participants rate the frequency and severity of the negative consequences they experienced due to alcohol use. The response options for each item range from 0 (never) to 4 (almost always), with some items having additional response options. The total score is the sum of all 50 items, with higher scores indicating more severe negative consequences related to alcohol use. The possible score on the DrInc scale ranges from 0 (no negative consequences) to 200 (highest score on all 50 items).
Symptom Checklist (SCL-90-R) | The questionnaire will be completed at screening (visit 1, approx. 14 days prior to the IMP-administration), and following IMP administration (approx. 28 days post-treatment and follow-ups)
  The "Symptom Checklist (SCL-90-R)" is a self-report inventory that assesses a broad range of psychological symptoms and psychological distress. It consists of 90 items that evaluate 9 domains of symptoms: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. The questions use a Likert scale, where participants rate the severity of symptoms they have experienced in the past week. The response options range from 0 (not at all) to 4 (extremely), with higher scores indicating more severe psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Preller, Dr., Principal Investigator — Psychiatric University Clinic
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rieser NM, Bitar R, Halm S, Rossgoderer C, Gubser LP, Thevenaz M, Kreis Y, von Rotz R, Nordt C, Visentini M, Moujaes F, Engeli EJE, Ort A, Seifritz E, Vollenweider FX, Herdener M, Preller KH. Psilocybin-assisted therapy for relapse prevention in alcohol use disorder: a phase 2 randomized clinical trial. EClinicalMedicine. 2025 Mar 14;82:103149. doi: 10.1016/j.eclinm.2025.103149. eCollection 2025 Apr. PMID 40144690